CLINICAL TRIAL: NCT06402266
Title: Effects of Transcranial Direct Current Brain Stimulation on Apolipoprotein-ε4 Allele Gene Carriers on an App-based Short-term Memory Task
Brief Title: Simultaneous tDCS and Computerised Gamified Short-term Memory Task Feasibility
Acronym: ACTTDCS-FG
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Brain+ ApS (Unknown); Eurostars EUREKA (Unknown); Innovation Fund Denmark (Individual)
Responsible Party: Sponsor
Other Study IDs: ACTTDCS
Record Dates: First submitted 2024-02-29; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-02

CONDITIONS: Genetic Predisposition
Keywords: Apolipoprotein E4; Cognitive reserve; Gamified cognitive training; Brain stimulation; tDCS; Technical compatibility
MeSH Terms: conditions — Genetic Predisposition to Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: tDCS — The STM task will be combined with respectively two times active tDCS and one sham tDCS. The 3 conditions will be randomised, and both scientific staff and participants will be blinded.
  Participants will perform the STM task on a tablet for 45 min. Headsets will deliver the tDCS. Two different placements will be used for the active stimulations: 1) F3 and PZ, and 2) F4 and PZ. The current output range will be 1.6mA and the stimulation will last for 30 min. The sham stimulation will function as a control condition. During the sham stimulation, the current density will be ramped up for 15 sec until the current reaches a density of 1.6mA for 60 sec and then again ramped down for 15 sec.
  After the session, participants will fill out a brief questionnaire regarding their experience.
  The time interval between sessions will be 1-3 weeks.

SUMMARY:
The goal of this observational study is to gain insight into the effects of transcranial direct current stimulation (tDCS) on short-term memory task performance and the feasibility of tDCS in overtly healthy carriers of the susceptibility allele, Apolipoprotein (APOE) ε4, for late-onset Alzheimers disease.

The main questions the study aims to answer are:

* If tDCS is feasible in overtly healthy APOE ε4 carriers using a headset and an app-based short-term memory task.
* If overtly healthy APOE ε4 carriers perform better on a complex short-term memory task when receiving tDCS to the right hemisphere (F4 à PZ) compared to the left hemisphere (F3 à PZ) or sham tDCS.

Participants will be asked to complete an app-based short-term memory task while receiving either tDCS to either the right or left hemisphere or sham stimulation on 3 different days spread out over 1-3 weeks.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common neurodegenerative disorder causing dementia. The most common form of AD is that of idiopathic AD, or late-onset AD, which typically affects individuals above the age of 65. Individuals, who are carriers of the Apolipoprotein (APOE) ε4 allele have an increased risk of developing late-onset AD, and AD brain pathology has been observed in APOE ε4 carriers as young as 55 years of age.

AD can be perceived as a continuum, with the pathophysiological disease process beginning in the brain many years prior to the onset of overt symptoms. Thus, individuals may show evidence of AD biomarkers in blood or cerebrospinal fluid or on brain scans in the absence of any overt symptoms. Individuals with incipient AD brain pathology but no overt symptoms may be classified as 'preclinical AD'. APOE ε4 allele carriage increases the risk of developing AD brain pathology 2-4 fold.

One of the most common cognitive symptoms in AD is memory impairment, such as impairments in short-term memory (STM). Subtle impairments in memory, including in STM, can even be detected in preclinical AD using sensitive memory tests. Therefore, STM may provide a suitable target to help preserve individual's cognitive functioning earlier in the disease process.

Cognitive reserve is a hypothetical construct proposed to explain the incongruency between the burden of AD pathology and cognitive dysfunction observed in some older individuals and has been defined as the ability to optimise or maximise performance through differential recruitment of brain networks. Epidemiological studies suggest that the cognitive reserve is increased by lifetime exposures, including educational and occupational attainment as well as leisure activities in late life. An underlying assumption is that these exposures improve brain plasticity. Cognitive training has shown positive effects with regards to promoting brain plasticity in older adults and could thus have the potential to foster or strengthen cognitive reserve in individuals at risk for developing AD later in life.

Cognitive training in combination with other neuroplasticity-enhancing techniques has been suggested as an option for promoting the positive effects of cognitive training alone. Transcranial direct current stimulation (tDCS) is a noninvasive neuro-modulatory technique where low intensity direct current is delivered to cortical areas to facilitate or inhibit ongoing, spontaneous neuronal activity. As tDCS has been shown to improve STM in healthy elderly participants, combining cognitive training with tDCS may be a way to enhance the effects of cognitive training and enhance cognitive reserve. Thus, it is sensible to explore the feasibility of tDCS on improving STM during a computerised game targeting STM, starting with healthy elderly APOE ε4 allele carriers, i.e. healthy elderly individuals, who are genetically predispositioned to AD, but who are otherwise healthy.

This study aims to investigate the effect of tDCS on memory performance on an app-based STM task in healthy elderly APOE ε4 carriers aged 55-75. All participants will be recruited from an existing in-house registry of individuals who have already been confirmed to be APOE ε4 carriers on a blood test. The tDCS or sham stimulation will be delivered by a headseat, where the spatial arrangement of the electrodes that delivers the stimulation and their outlets used in the stimulation determines the regions and distributed networks of the brain being stimulated. Participants will first try out the app-based STM task on its own in order to become familiar with it. Thereafter, they will come in on 3 different days within 1-3 weeks, where they will complete the same STM task again while undergoing either active or sham tDCS. This will allow for the examination of whether active tDCS can improve memory performance on this type of complex STM task in overall healthy elderly individuals who are genetically predisposed for late-onset AD.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 55-75 years old
* The participant is confirmed to carry at least one APOE ε4 allele on a blood test
* The participant has at least 7 years of education or a good working history
* Normal cognition (MMSE score > 26)

Exclusion Criteria:

* Any dementia
* Significant systematic disease
* Severe and unstable medical disease or psychiatric disorder, including medications for these diseases or disorders
* Past history of stroke or brain damage
* Epilepsy or history of epileptic seizures
* Migraine
* Skin or scalp condition in the areas where the electrodes will be placed
* Depression
* Alcohol or drug abuse
* Significantly impaired vision or hearing
* Colour blindness
* Adverse effects to previous tDCS or other brain stimulation techniques

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthy elderly APOE ε4 carriers recruited from an existing, in-house registry.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Observations of the feasibility of simultaneous tDCS with a computerised, gamified short-term memory task | During stimulation (up to 1 hour)
  The first outcome measure has to do with whether it is feasible to deliver tDCS via a portable headset while participants perform a computerised gamified STM task, in order to evaluate whether this would be possible in a home-based setting. This will be measured is by observing the sessions with this set-up and noting down difficulties during the session, including technical challenges and participant complaints.
Participants' self-reported experience of the simultaneous tDCS with a computerised, gamified short-term memory task assessed by a self-report questionnaire | Post-stimulation (through study completion, up to 1 year)
  The second outcome measure has to do with how the participants experienced the session. This will be assessed by having participants answer a self-report questionnaire on their experience after the session. The questionnaire consists of 3 overarching questions: 1) how the participants felt wearing the head-set; 2) how they experienced the stimulation, including whether they felt any discomfort; and 3) and how they experienced the overall set-up with the headset and the gamified STM task, including their assessment on whether they think it will work in a home-based setting.
Effects of tDCS on computerised gamified short-term memory task performance | Post-stimulation (through study completion, up to 1 year)
  The third outcome measure has to do with whether simultaneous brain stimulation affects participants' performance on the gamified STM task; or, more specifically, whether participants receiving tDCS stimulation performed better than those receiving sham stimulation. This is done by automatically logging the task data, which can then be accessed after the session. The outcome is evaluated as one overall score of STM performance based upon 1) identification accuracy, and 2) placement accuracy. A higher overall STM performance score indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob U Blicher, Assoc. Prof., Principal Investigator — Aarhus University, Centre for Functionally Integrative Neuroscience (CFIN)
Locations (1):
- Aarhus University, Centre for Functionally Integrative Neuroscience, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-09-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT06402266/ICF_000.pdf